CLINICAL TRIAL: NCT07279831
Title: Brain-lung Interactions in Patients Receiving High-flow Humidified Oxygen for de Novo Acute Hypoxemic Respiratory Failure
Brief Title: Brain-lung Interaction During Acute Respiratory Failure
Acronym: BrainFlow
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251258
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; High flow nasal cannulae; Electroencephalogram; Near infrared spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients admitted to critical care for acute renal failure
  Interventions: Diagnostic Test: EEG/NIRS/EMG

INTERVENTIONS:
Diagnostic Test: EEG/NIRS/EMG — Two 10-minute recordings will be made. Each recording will include continuous collection of EEG, NIRS, and EMG data from the scalene muscles, as well as collection of intensive care monitoring variables every minute.

SUMMARY:
Acute hypoxemic de novo respiratory failure (AHRF) is a common cause of admission to the intensive care unit (ICU). Its main cause is community-acquired pneumonia. Prevention of intubation relies, among other things, on high-flow nasal canulae (HFNC). However, approximately 40% of patients are intubated despite HFNC.

Our team has developed measurements derived from electroencephalograms (EEG) and near-infrared spectroscopy (NIRS) that enable the study of brain-ventilation interactions. To date, these tools have been studied exclusively in intubated patients. the investigators now wish to study them in non-intubated patients.

The objective of this study is to investigate the relationship between the brain and lungs in adult patients admitted to the intensive care unit for acute hypoxemic respiratory failure and for whom the attending physician has decided to initiate HFNC.

Before and one hour after the introduction of HFNC, electroencephalogram (EEG), near-infrared spectroscopy (NIRS), and electromyogram (EMG) of the Scalen muscles will be collected.

From these recordings, the following variables will be collected: 1) The density of the gamma (30-100 Hz), beta (13-30 Hz), alpha (8-12 Hz), theta (4-8 Hz), and delta (0.5-4 Hz) frequency spectrum of the EEG in each of the following right and left cortical regions: medial region of the prefrontal cortex, anterior region of the cingulate gyrus, posterior region of the cingulate gyrus, insula, somatosensory cortex, angular gyrus, lateral prefrontal cortex, and supplementary motor area; 2) Connectivity between these regions for each frequency spectrum; 3) Pre-inspiratory potential; 4) Rieman classifier; 5) Coherence and Granger causality between each frequency spectrum and the scalene muscles EMG.

These variables will be compared before and 1 hour after initiation of HFNC and between patients who will be intubated because of HFNC failure and those who will not.

DETAILED DESCRIPTION:
Acute hypoxemic de novo respiratory failure (AHRF) is a common cause of admission to the intensive care unit (ICU). Its main cause is community-acquired pneumonia. Prevention of intubation relies, among other things, on high-flow nasal canulae (HFNC). However, approximately 40% of patients are intubated despite HFNC.

Our team has developed measurements derived from electroencephalograms (EEG) and near-infrared spectroscopy (NIRS) that enable the study of brain-ventilation interactions. To date, these tools have been studied exclusively in intubated patients. the investigators now wish to study them in non-intubated patients.

The objective of this study is to investigate the relationship between the brain and lungs in adult patients admitted to the intensive care unit for acute hypoxemic respiratory failure and for whom the attending physician has decided to initiate HFNC.

Before and one hour after the introduction of HFNC, electroencephalogram (EEG), near-infrared spectroscopy (NIRS), and electromyogram (EMG) of the Scalen muscles will be collected.

From these recordings, the following variables will be collected: 1) The density of the gamma (30-100 Hz), beta (13-30 Hz), alpha (8-12 Hz), theta (4-8 Hz), and delta (0.5-4 Hz) frequency spectrum of the EEG in each of the following right and left cortical regions: medial region of the prefrontal cortex, anterior region of the cingulate gyrus, posterior region of the cingulate gyrus, insula, somatosensory cortex, angular gyrus, lateral prefrontal cortex, and supplementary motor area; 2) Connectivity between these regions for each frequency spectrum; 3) Pre-inspiratory potential; 4) Rieman classifier; 5) Coherence and Granger causality between each frequency spectrum and the scalene muscles EMG.

These variables will be compared before and 1 hour after initiation of HFNC and between patients who will be intubated because of HFNC failure and those who will not.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* Admitted to the intensive care within the last 48 hours
* De novo acute hypoxemic respiratory failure with an indication for high-flow nasal cannula (HFNC), defined by the combination of the following three criteria:

  * Tachypnea > 25 breaths/min or labored breathing
  * PaO2 (partial pressure of oxygen ) /FiO2 ( fraction of inspired oxygen ) ≤ 200 mmHg
  * Unilateral or bilateral alveolar opacities on chest X-ray
* Decision by the attending physician to initiate HFNC treatment
* After information, the patient or next of kind did not refuse to participate (according to the French law, written informed consent is waived)

Exclusion Criteria:

* - Exacerbation of an underlying chronic respiratory disease
* Acute cardiogenic pulmonary edema indicating non-invasive ventilation (NIV)
* Hypercapnia > 45 mmHg indicating NIV
* Glasgow Coma Scale < 13
* Imminent intubation
* Underlying central neurological disease likely to alter EEG signals
* Pregnancy or breastfeeding
* Lack of health insurance coverage
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to critical care for acute renal failure
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
density of the gamma frequency spectrum of the EEG in the medial region of the right prefrontal cerebral cortex | before and 1 hour after initiation of high flow nasal cannulae
  density of the gamma frequency spectrum (30 - 100 Hz) of the EEG in the medial region of the right prefrontal cerebral cortex, before initiation of HFO ( = high-flow oxygen), then 1 hour after its initiation

SECONDARY OUTCOMES:
The density of the gamma, beta, alpha, theta, and delta frequency spectrum | before and 1 hour after initiation of high flow nasal cannulae
  The density of the gamma frequency spectrum (30-100 Hz) of the EEG in the following cortical regions: medial region of the left prefrontal cortex, anterior region of the right and left cingulate gyrus, posterior region of the right and left cingulate gyrus, right and left insula, right and left somatosensory cortex, right and left angular gyrus, right and left lateral prefrontal cortex, and right and left supplementary motor area. and the densities of the beta (13-30 Hz), alpha (8-12 Hz), theta (4-8 Hz), and delta (0.5-4 Hz) frequency spectra in each of the aforementioned right and left cortical regions.
Connectivity | before and 1 hour after initiation of high flow nasal cannulae
  Connectivity between the medial region of the prefrontal cerebral cortex, the anterior region of the cingulate gyrus, the posterior region of the cingulate gyrus, the insula, the medial region of the prefrontal cortex, the somatosensory cortex, the angular gyrus, the lateral prefrontal cortex and the supplementary motor area, right and left, for the gamma (30-100 Hz), beta (13-30 Hz), right and left, alpha (8-12 Hz), right and left, theta (4-8 Hz) and delta (0.5-4 Hz), right and left frequency spectra.
pre-inspiratory potential | before and 1 hour after initiation of high flow nasal cannulae
  the presence of a pre-inspiratory potential will be searched for
Riemann classifier | before and 1 hour after initiation of high flow nasal cannulae
  The area under the curve of the receiver operating characteristics (ROC) of the Riemann classifier will be measured.
Coherence and Granger Causality | before and 1 hour after initiation of high flow nasal cannulae
  The coherence between the EMG and the EEG frequency bands gamma (30-100 Hz), beta (13-30 Hz), right and left, alpha (8-12 Hz), theta (4-8 Hz), and delta (0.5-4 Hz), right and left. If significant coherence exists, the direction of the relationship is determined using Granger causality.
Oxyhemoglobin (HbO2) concentration | before and 1 hour after initiation of high flow nasal cannulae
  Oxyhemoglobin (HbO2) concentration derived from optical densities (fNIRS) using the modified Beer-Lambert law, in the prefrontal and lateral regions of the cortex, right and left.
Change in amplitude for fNIRS frequencies (fNIRS) | before and 1 hour after initiation of high flow nasal cannulae
  The change in amplitude for frequencies (fNIRS) between 1.0 and 1.25 Hz (related to heart rate), between 0.18 and 0.25 Hz (related to respiratory rate), between 0.08 and 0.13 Hz (related to myogenic frequency, sympathetic tone), between 0.05 and 0.07 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, Principal Investigator — APHP
Locations (1):
- Service de Médecine Intensive et Réanimation, Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.